CLINICAL TRIAL: NCT00405119
Title: A Randomized, Double-blind, Four Period Cross-over Comparison of the Effect of Two Doses Lavoltidine, Esomeprazole, and Placebo on 24 Hour Gastric pH and Frequency of Heartburn in Symptomatic GERD Subjects Without Esophageal Erosions
Brief Title: A Study To Investigate The Effectiveness Of AH234844 (Lavoltidine) Compared With NEXIUM And Ranitidine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: LAV104616
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Gastroesophageal Reflux Disease; Reflux, Gastroesophageal
Keywords: tolerance; pharmacodynamics; ranitidine; esomeprazole; pharmacokinetics; gastroesophageal reflux disease (GERD); AH23844
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — loxtidine; Esomeprazole; Ranitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AH23844 (lavoltidine)
Drug: NEXIUM (esomeprazole)
Drug: ZANTAC (ranitidine)
  Other Names: AH23844 (lavoltidine); NEXIUM (esomeprazole)

SUMMARY:
Current treatment for gastroesophageal reflux disease (GERD) confirms an unmet need in patients, based on slow onset of action and an inability to provide 24-hour gastric-acid suppression. Clinical data on AH234844 demonstrates a rapid onset of action, high potency, and prolonged duration of effect. The present study endeavors, in part, to compare lavoltidine to two GERD drugs, NEXIUM and ranitidine.

DETAILED DESCRIPTION:
A three-part study in healthy male volunteers to determine the most effective of four different lavoltidine doses on gastric pH and to compare the most effective dose with NEXIUM (esomeprazole) 40mg for the inhibition of gastric-acid secretion and with ranitidine (300mg/day) for the amount of pharmacodynamic tolerance

ELIGIBILITY:
Inclusion criteria:

* Subject must have a Body Mass Index (BMI) from 19-30 kg/m2
* Subject does not present with abnormal clinical lab findings
* Subject is able to tolerate a nasogastric pH electrode.

Exclusion criteria:

* Subject is Helicobacter-positive on a C13 urea breath test
* Subject has a baseline median 24-hour gastric pH>3
* For Part B of the study, subjects are CYP 2C19 poor metabolizers.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
pH over 24hours | over 24hours

SECONDARY OUTCOMES:
%24 hours pH>4 Median gastric pH Adverse events | over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Herston, Queensland